CLINICAL TRIAL: NCT01147562
Title: Biomarker Discovery and Validation in Lung Cancer
Acronym: LCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Guy Berchem (Other)
Collaborators: Integrated Biobank of Luxembourg (Other); Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor-Investigator, Dr. Guy Berchem, MD, Public Research Centre Health, Luxembourg
Organization: Public Research Centre Health, Luxembourg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IBBL0001
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Biopsy; Biomarker; Tissue Collection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung Cancer Patients (Other): Patients with a suspected or confirmed diagnosis of lung cancer, whether or not scheduled for lesion biopsy, thoracentesis or surgical resection of their tumor
  Interventions: Procedure: Collection of biospecimen

INTERVENTIONS:
Procedure: Collection of biospecimen — Collection of saliva, blood and tissues from subjects diagnosed with lung cancer, who are scheduled for biopsy of their lesion or surgical resection of their tumor.

SUMMARY:
Lung cancer is responsible for the most deaths due to cancer each year in both men and women worldwide and once diagnosed, the 10 year survival rate is poor (<15%). This poor prognosis is based in large part on the absence of an effective diagnostic test for the disease. The chief objective of this study is to develop a molecular-based diagnostic test specific for lung cancer. Subjects suspected or diagnosed with lung cancers, who are either undergoing thoracentesis, biopsy of a suspicious lesion or surgical resection of their tumor will be asked to participate in this study. Those subjects, who will undergo surgical resection, will donate both lung tumor tissue and adjacent normal lung tissue (potentially including lymph nodes), while non-surgical candidates will donate a portion of their excess biopsy sample, if available, after diagnosis has been confirmed. Subjects undergoing thoracentesis for pleural effusion will donate a portion of their fluid sample, if the fluid volume collected is in excess of that needed for clinical care purposes. Blood samples and optionally saliva will also be collected from all subjects, whether undergoing surgery or not. In addition to biosample collection, detailed annotated demographic and clinical information will be collected from subjects. Subjects will be followed for outcome analysis, specifically for tumor recurrence, every 6 months, during 5 years. In case of change in chemotherapy treatment, biosamples and clinical information will also be collected. Collected biosamples will be analyzed using a series of molecular and proteomic technologies for developing biomarkers of the disease.

DETAILED DESCRIPTION:
The primary objective of this study is to discover and validate molecular biomarkers for lung cancer.

Lung cancer remains the leading cause of cancer death in industrialized countries. Most patients with non-small cell lung cancer (NSCLC) present with advanced disease, and despite recent advances in multi-modality therapy, the overall 10-year survival rate is less than 10%. A significant minority of patients (25-30%) with NSCLC have stage I disease and receive surgical intervention alone. Although 35-50% of patients with stage I disease will relapse within 5 years, it is not currently possible to identify specific high-risk patients. In addition, for patients with metastatic disease, standard chemotherapeutic approaches result in less than 50% response rate, meaning that more than half of patients do not benefit and only suffer from side effects.

Only very limited data exists on markers capable of predicting response to chemotherapy.

This population would certainly also benefit from more of those markers. Another situation where a biomarker could be potentially very useful is the situation where a pulmonary nodule is diagnosed and has to be characterized. In this situation a biomarker could predict whether the nodule is or is not cancerous and thus, make CT Scan follow up unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspected or confirmed diagnosis of lung cancer, whether or not scheduled for lesion biopsy, thoracentesis or surgical resection of their tumor

Exclusion Criteria:

* Pregnant women
* Minors (subjects less than 18 years of age)
* Prisoners
* Subjects unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-10-14 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Discover and validate molecular biomarkers for lung cancer | Participants are followed up very 6 months up to to 5 years or until death.
  Investigate markers capable of prediciting response to chemotherapy. In cas a pulmonary nodule is diagnosed and has to be characterized, a biomarker could predict whether the nodule is or is not cancerous and thus, make CT Scan follow up unnecessary.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Berchem, MD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (2):
- Luxembourg (2):
  - Centre Hospitalier de Luxembourg (CHL), Luxembourg
  - Clinique Sainte Thérèse (Zithaklinik), Luxembourg

REFERENCES:
- [Background] Dziadziuszko R, Hirsch FR. Advances in genomic and proteomic studies of non-small-cell lung cancer: clinical and translational research perspective. Clin Lung Cancer. 2008 Mar;9(2):78-84. doi: 10.3816/CLC.2008.n.012. PMID 18501093
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875